CLINICAL TRIAL: NCT02887664
Title: The Correlation Between the n-6:n-3 Ratio and Inflammatory Markers in Small for Gestational Age (SGA) Infants Compared With Appropriate for Gestational Age (AGA) Infants
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0285-16-TLV-DM
Record Dates: First submitted 2016-08-22; First posted 2016-09-02 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Small for Gestational Age Infants; Appropriate for Gestational Age Infants
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Blood test in Mothers of SGA Infants: In mothers of Small for Gestational Age (SGA) Infants, maternal and cord blood test will be performed
  Interventions: Procedure: Blood test
- Blood test in Mothers of AGA infants: In mothers of Appropriate for Gestational Age (AGA) Infants, maternal and cord blood test will be performed
  Interventions: Procedure: Blood test

INTERVENTIONS:
Procedure: Blood test — Blood will be drawn from mother's vein and from the cord to test for n-6:n-3 ratio and inflammatory markers: CRP, IL-6, TPO and TNF-alpha markers

SUMMARY:
Numerous studies have recommended the use of n-3 PUFA supplementation during human pregnancy and lactation for the prevention of preterm birth, beneficial effects on fetal development, visual and cognitive development and other functional outcomes of the infants.

The aim of the present study is to assess the correlation between ratio of n-3:n-6 fatty acid and inflammation markers in SGA infants compared with appropriate for gestational age (AGA) infants. The investigators hypothesize that in SGA infants n-3 and n-6 fatty acid concentrations in cord blood will differ from those observed in AGA and might correlate with the level of circulating mediators.

ELIGIBILITY:
Inclusion Criteria:

* Mothers of SGA infants ( above 35 week of gestation)
* Mothers of term and near-term AGA infants

Exclusion Criteria:

* Maternal chronic diseases, smoking, diabetes, alcohol use, pregnancy-associated hypertension and pre-eclampsia
* Neonatal depression
* Congenital malformations
* Intrauterine infections
* Chromosomal aberrations
* Mothers interested in cord blood banking

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Mothers of term or or near term infants after delivery
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-10-02 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Cord blood analysis | at time of delivery
  Determination of the cord blood values of inflammatory markers (CRP, IL-6, TPO, TNF-alpha) and of the n-6:n-3 ratio

SECONDARY OUTCOMES:
Maternal blood analysis | at time of delivery
  Determination of the maternal blood values of inflammatory markers (CRP, IL-6, TPO, TNF-alpha) and of n-6:n-3 ratio

CONTACTS AND LOCATIONS:
Overall Officials: Dror Mandel, MD, Principal Investigator — Department of Neonatology, Lis Maternity Hospital, Tel Aviv Medical Center
Locations (1):
- Sourasky medical center (Ichilov), Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No